CLINICAL TRIAL: NCT06526390
Title: Flexible Ureteroscopy With Tip-Bendable Suction Ureteral Access Sheath Versus Mini-Percutaneous Nephrolithotomy for Treatment of 2-3cm Renal Stones: an International Multicentre, Randomized, Parallel-Group, Non-Inferiority Trial
Brief Title: Flexible Ureteroscopy With Tip-bendable Suction Ureteral Access Sheath Versus Mini-Percutaneous Nephrolithotomy for Treatment of 2-3cm Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: University of Malaya (Other); Ankara University (Other); Saint Petersburg State University Hospital (Unknown); Fortune Urology Clinic (Unknown); Guizhou Provincial People's Hospital (Other); Baoshan No.2 People's Hospital (Unknown); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shengjing Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MERE2024-001
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Urolithiasis; Kidney Stone
Keywords: kidney stone; Flexible ureteroscopy; PCNL
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients and surgeons cannot be blinded to the allocated trial arm due to the differing nature of the interventions. However, the radiologists assessing the post-operative imaging (CT scans) will be blinded to the intervention. The postoperative clinical assessment will be performed by investigators who are blinded to the surgical procedures and had not been involved in the surgeries. We will perform blinded statistical analyses, in which the individual performing the analyses in unaware the group belonging. The code for group assignment will not be broken until the analyses and interpretation have been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- f-URS with S-UAS group (Experimental): f-URS with S-UAS will be performed for patients.
  Interventions: Procedure: f-URS
- mini-PCNL group (Other): mini-PCNL will be performed for patients.
  Interventions: Procedure: mini-PCNL

INTERVENTIONS:
Procedure: f-URS — f-URS with S-UAS
  Arms: f-URS with S-UAS group
Procedure: mini-PCNL — mini-PCNL
  Arms: mini-PCNL group

SUMMARY:
Background: Percutaneous nephrolithotomy (PCNL) is the first-line treatment for renal stones larger than 2 cm according to EAU and AUA guidelines. Advances in flexible ureteroscopy, including smaller disposable ureteroscopes and suction techniques, have expanded its indications. The tip-bendable suction ureteral access sheath (S-UAS) offers improved flexibility and stone-free rates (SFR). This study compares clinical outcomes of flexible ureteroscopy (f-URS) with S-UAS and mini-PCNL in treating 2-3 cm renal stones.

Objective: This study aims to determine if f-URS with S-UAS is non-inferior to mini-PCNL regarding stone-free rates. Secondary objectives include comparing complication rates, surgical time, and hospitalization duration.

Methods: This multicenter, international, prospective, non-inferiority, randomized controlled trial will enroll 720 patients across 12 urological centers. Patients will be randomized to either f-URS with S-UAS or mini-PCNL. Outcomes include immediate and 3-month SFR, operative time, hospital stay, further interventions, complications, and quality of life.

Results: Data will be analyzed using intention-to-treat and per-protocol approaches, with statistical analyses performed using SPSS software.

Conclusion: This study will provide high-level evidence on the effectiveness of f-URS with S-UAS compared to mini-PCNL for medium-sized renal stones.

DETAILED DESCRIPTION:
1. Background

   According to the EAU and AUA guidelines, percutaneous nephrolithomy (PCNL) remains the first-line treatment for renal stones larger than 2 cm. In recent years, advancement in flexible ureteroscopic technology, such as the emergence of smaller disposable flexible ureteroscopes and suction techniques, have increased the efficiency of flexible ureteroscopy and expanded its indications.

   The tip bendable suction ureteral access sheath (S-UAS) is a novel UAS characterized by excellent flexibility and bendability at the tip, enabling passive bending (angle >90°) in sync with the bending of flexible ureteroscope. It can be connected to a vacuum suction device. Initial studies suggest that S-UAS can significantly improve stone-free rates (SFR) and reduce the complication rates. Given the significant improvements in the effectiveness of flexible ureteroscopy (f-URS) with S-UAS, several studies report favorable outcomes in managing renal stones ≥2cm using flexible ureteroscopy. However, high-level evidence is still lacking to determine whether flexible ureteroscopy with S-UAS can achieve outcomes comparable to PCNL for medium-sized stones (2-3cm).

   The objective of the current study is to assess the clinical outcomes of f-URS with S-UAS and mini-PCNL in the treatment of 2-3 cm renal stones, aiming to evaluate the suitability of f-URS for these patients.
2. Study objectives

   The aim of this study is to determine whether f-URS with S-UAS is non-inferior to mini-PCNL in terms of surgical efficiency for 2-3 cm renal stones. An initial pilot phase will be included to assess the feasibility of recruitment and the appropriateness of eligibility criteria and outcome measures. The research question to be addressed is: does f-URS with S-UAS result in non-inferior stone-free rates compared to mini-PCNL? The secondary objective is to compare the complication rates, surgical time, and hospitalization time.
3. Methods and Design

This trial is a multicentre, international, prospective, parallel-group, non-inferiority, randomized, controlled trial.

3.1 Study overview

This trial is a multicentre, international, prospective, parallel group, non-inferiority, randomized, controlled trial.

3.2 Setting

The study will be conducted across 12 urological departments with a notable caseload of urinary stones (8 in China, one in Malaysia, one in Russian Federation, one in India and one in Turkey). Each participating center routinely performs over 300 f-URS and 100 mini-PCNL procedures annually.

3.3 Population

Inclusion criteria:

1. Adults aged ≥ 18 years;
2. American Society of Anesthesiology score 1-3;
3. Renal stones diameter of 2-3 cm confirmed by non contrast-CT;
4. Capable of giving written informed consent, including adherence to the requirements of the trial.

Exclusion criteria:

1. Patients with abnormal urinary tract anatomy (such as horseshoe kidney or ileal conduit);
2. Patients with uncontrolled urinary tract infection;
3. Patients with health or other factors that are absolute contraindications to f-URS or mini-PCNL;
4. Patients unable to understand or complete trial documentation.

3.4 Identification and Enrolment of potential participants

Local procedures at participating hospitals may vary; therefore, the timing and mode of approach to patients and the consent process will be adapted to accommodate both site variability and patient needs. As standard practice, clinicians or delegated personnel will assess patients presenting with suspected renal stones. A log will be maintained of all patients assessed to document reasons for non-inclusion in the study (e.g. reason for ineligibility or refusal to participate) to inform the CONSORT diagram. Brief details of potentially eligible patients will be recorded in the screening logs at each site to aid in monitoring potential participant inclusion.

Following confirmation of renal stones by CT scan, eligible patients (according to the inclusion and exclusion criteria) will be provided with a patient information leaflet. This leaflet will inform them of the benefits and known drawbacks of all aspects of this trial. The patient information leaflet explains that the trial is investigating the use of either f-URS or mini-PCNL as the treatment option for renal stones. Each patient will have the opportunity to discuss the study with the local clinical team. Patients may decide to participate during a consultation with the local clinical team, either during a clinic appointment or while hospitalized for their initial stone episode.

Signed informed consent forms will be obtained from the participants at all centres. Participants who cannot give informed consent (e.g. due to incapacity) will not be eligible for participation. The participant's permission will be sought to inform their general practitioner that they are taking part in this trial. Participants will be randomized to one of the two groups following consent, and completion of baseline questionnaire.

3.5 Randomization and allocation

Randomization will be conducted using a stratified approach based on the participating centers. Each center of the 12 centers will enroll 60 participants, Participants within each center will be randomized to either the f-URS group or the mini-PCNL group in a 1:1 ratio. Randomization sequence generation will be performed electronically before patient participation. Random sequence allocation and concealment will be implemented using consecutively numbered, sealed envelopes. When the patient has signed the informed consent form and the decision for surgery has been made, the envelope will be opened to determine the surgical method.

3.6 Intervention

Two interventions will be evaluated: (1) f-URS with S-UAS and (2) mini-PCNL.

3.7 Operation protocol

A standardized operating methodology, authorized by the principal investigator at each center, will be established and endorsed to ensure consistency. Monthly protocol monitoring visits will be carried out across all participating centers to guarantee adherence to the established procedures.

A non-contrast CT scan with a 2-mm thickness will be routinely performed to determine the location and size of the stone (including stone diameter, stone area, and stone volume). Stone burden and density will be consistently measured using identical software across all centers. All patients will receive standard peri-operative antibiotic prophylaxis (a single dose of cefuroxime 1500 mg or levofloxacin 500 mg in cases of allergy, depending on the respective center's standard practice protocol) administered 0.5 hours before the intervention. Patients with a positive preoperative urine culture will be treated with appropriate antibiotics based on the culture sensitivity results for 4-7 days prior to the operation.

Endoscopic procedure

f-URS

The procedure will be performed under general anesthesia, and the lithotomy position will be adopted for each procedure. A 5 Fr open-ended ureteral catheter will be inserted into the ureter, and retrograde pyelography (RPG) will be performed to assess the upper urinary tract. Subsequently, a 0.035/0.038-inch guidewire will be placed into the renal pelvis. Either a 12/14 Fr or 11/13 Fr S-UAS will be utilized. In cases where the UAS cannot be placed due to a narrow ureter, a smaller UAS (10/12 Fr) will be attempted. If a 10/12 Fr UAS cannot be successfully placed, a double-J stent will be left in situ, and the procedure will be terminated. The second-session f-URS will be performed 2 weeks after the placement of the double-J stent.

f-URS will be performed using two types of digital flexible ureteroscopes: 8.5Fr and 7.5Fr. Either an 8.5 Fr or 7.5 Fr disposable flexible ureteroscope will be selected for the f-URS based on the UAS size: an 8.5 F scope for 12/14 F UAS, and a 7.5 F scope for 11/13 F or 10/12 F UAS.

The stone will be fragmented by a holmium laser (Ho:YAG) or Thulium Fiber laser (TFL), using a 200 µm laser fiber with an energy setting less than 30 W. An irrigation pressure pump will be utilized, with the irrigation flow rate will be set at 50-100 ml/min. The suction pressure will be controlled to a setting of 80-120 mmHg. At the end of each procedure, the UAS will be removed along with the ureteroscope.

A 6 Fr indwelling double-J stent will be placed post-operatively and kept for 2 weeks, depending on the condition of the ureter. A postoperative Foley catheter will not be placed routinely.

Mini-PCNL

Under general anesthesia, a 5 Fr ureteral catheter will be inserted into the target ureter using a ureteroscope, and the bladder will be drained with a 16 Fr Foley catheter. The patient will then be turned to the prone position. Percutaneous access will be achieved using an 18-gauge coaxial needle to puncture the desired calyx under fluoroscopic or ultrasound guidance. Tract dilatation will be accomplished using fascial dilators up to 18 Fr. When multiple nephrostomy tracts are necessary to remove the stones, the same technique will be employed for each tract. Fragmentation of the stone burden will be accomplished using either a pneumatic lithotripter, holmium laser (Ho:YAG) or Thulium Fiber laser (TFL). At the end of the procedure, a 6 Fr double-J ureteral stent will be left in place. The decision to leave a silastic nephrostomy tube will be depending on the clinical decision of each operating surgeon.

3.8 Follow-up and data collection

Low-dose non-contrasted CT, with a 2-mm section thickness will be performed within 72 hours postoperatively to assess immediate SFR. SFR is defined as no residual stone visualized under endoscopy and absence of fragments in the kidney or fragments ≤ 2 mm. Blood routine examination and serum procalcitonin will be performed within 2 hours after the operation to monitor for infection. Haemoglobin decrease will be documented by comparing the preoperative value to that 24-h postoperatively. Whole blood transfusion will be given for patients with postoperative haemoglobin of <80 g/L. For f-URS group, if experiencing no significant postoperative discomfort, will be discharged the day after surgery. For mini-PCNL group, if nephrostomy tube was inserted, it will be removed 1-3 days after the drainage become grossly clear, and the patients will then be discharge. The double-J stent will be removed 2 weeks after surgery. Quality of Life (QOL) Score will be evaluated preoperatively and one-month postoperatively. Stone composition will be analyzed using the same infrared spectrometer and methodology at all centers. Low-dose CT scans will be obtained for all patients at the 3-month follow-up to evaluate the final stone-free status.

Patients' characteristics and clinical outcomes will be meticulously recorded on a pre-established case report forms (CRFs). Stone size will be defined as the largest diameter for a single stone and the sum of the largest diameters for multiple stones. Stone size and Hounsfield Unit (HU) will be consistently measured using identical software across all centers. Hydronephrosis will be graded according to the Onen hydronephrosis grading system (updated 2016). Operative time will be defined as the duration from the insertion of the endoscope into the urethra to the completion of stent placement for f-URS group, and from the start of the start of the percutaneous puncture to completion of nephrostomy tube placement for the mini-PCNL group. Hospital stay will be rounded to the nearest whole day and calculated from the day of surgery to the day of discharge.

Four CRFs will be completed by the research team at the recruiting site. A baseline CRF at randomization, a treatment CRF post-intervention, and CRFs at 1 month and 3 months post-operation. These will include additional interventions received and complications.

3.9 Outcome measures

Primary outcome

Immediate stone-free rate (SFR): no residual stone visualized under endoscopy and no residual stone or stone fragments less than 2 mm on low dose CT scan with a 2-mm section thickness within postoperative 72 hours are defined as stone free.

Secondary outcomes

1. Final SFR: SFR at 3 months postoperative based on CT scans.
2. Operative time.
3. Duration of hospital stay: rounded to the nearest whole day and calculated from the day of surgery to the day of discharge.
4. Further interventions received up to 3 months post randomization.
5. Complications up to 3 months post randomization (according to the Clavien-Dindo grading system8).
6. Improvement of Quality of Life Score: recorded preoperatively and at one month postoperatively using Wisconsin Stone QoL questionnaire.

3.10 Blinding

Patients and surgeons cannot be blinded to the allocated trial arm due to the differing nature of the interventions. However, the radiologists assessing the post-operative imaging (CT scans) will be blinded to the intervention. The postoperative clinical assessment will be performed by investigators who are blinded to the surgical procedures and had not been involved in the surgeries. We will perform blinded statistical analyses, in which the individual performing the analyses in unaware the group belonging. The code for group assignment will not be broken until the analyses and interpretation have been completed.

3.11 Subject withdrawal

Participants will remain in the trial unless they chose to withdraw consent or if they are unable to continue for a clinical reason. If a participant withdraws consent, permission will be sought to continue collecting outcome data from their healthcare records. All other changes in status, except for formal withdrawal of consent, will mean the participant is still followed up for all study outcomes wherever possible.

3.12 Sample size

The original sample size calculations reflect that the trial is non-inferiority design. Preliminary data suggested that the immediately SFR in the mini-PCNL arm and f-URS arm will be about 85% for treating of 2-3 cm renal stones. The margin of inferiority deemed acceptable is 8%. The sample size was estimated using simulations run in Stata. With 80% power and alpha set at 2.5%, 313 participants per group (626 in total) are required. To account for patients lost to follow-up and study withdrawals, this number was increased to 360 per group (720 in total).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 years;
2. American Society of Anesthesiology score 1-3;
3. Renal stones diameter of 2-3 cm confirmed by non contrast-CT;
4. Capable of giving written informed consent, including adherence to the requirements of the trial.

Exclusion Criteria:

1. Patients with abnormal urinary tract anatomy (such as horseshoe kidney or ileal conduit);
2. Patients with uncontrolled urinary tract infection;
3. Patients with health or other factors that are absolute contraindications to f-URS or mini-PCNL;
4. Patients unable to understand or complete trial documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Immediately stone-free rate (SFR) | Up to 72 hours.
  No residual stone visualized under endoscopy and no residual stone or stone fragments less than 2 mm on low dose CT scan with a 2-mm section thickness within postoperative 72 hours are defined as stone free.

SECONDARY OUTCOMES:
Final SFR | 3 months.
  SFR at 3 months postoperative based on CT scans.
Operative time | through operation completion, an average of 1 hour
  Operative time.
Duration of hospital stay | Up to 3 months.
  Rounded to the nearest whole day and calculated from the day of surgery to the day of discharge.
Further interventions (Second-look PCNL or RIRS or SWL) | Up to 3 months.
  Further interventions
Complications | Up to 3 months.
  Complications
Improvement of Quality of Life Score | Up to 3 months.
  Improvement of Quality of Life Score

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Zhu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not share to other researchers as ethical issues.

REFERENCES:
- [Derived] Zhu W, Ann Chai C, Ma J, Ilker Gokce M, Gadzhiev N, Kalathia J, Jiang K, Duan X, Cao J, Wu R, Song R, Bai S, Li X, Liu S, Zeng G. Flexible Ureteroscopy with a Tip-bendable Suction Ureteral Access Sheath Versus Mini-Percutaneous Nephrolithotomy for Treatment of 2-3-cm Renal Stones: Study Protocol for an International, Multicenter, Randomized, Parallel-group, Noninferiority Trial. Eur Urol Open Sci. 2024 Nov 4;70:167-173. doi: 10.1016/j.euros.2024.10.014. eCollection 2024 Dec. PMID 39559532